CLINICAL TRIAL: NCT07212985
Title: Horizontal Anterior Maxillary Ridge Augmentation Using Autogenous Ring Block Grafts Combined With Particulate Xenogeneic Bone Versus Biphasic Beta-tri-calcium Phosphate Sulphate EthOss Graft: A Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Nora Abdelgawad Mohamed, Associate Professor of Oral Medicine, Periodontology and Diagnosis, Faculty of Dental Medicine for girls, Al -Azhar University, Cairo, Egypt, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-PD-24-22
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Implant Dentistry
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABG + Xenograft + Collagen Membrane (Experimental): Patients receive autogenous bone block graft (from chin) combined with particulate bovine xenograft (Bio-Oss, Geistlich Pharma AG) and covered with absorbable collagen membrane (Bio-Gide).
  Interventions: Procedure: Autogenous Bone Block + Xenograft + Collagen Membrane
- ABG + EthOss (Synthetic Graft) (Experimental): Patients receive autogenous bone block graft (from chin) combined with EthOss, a biphasic synthetic graft material (35% calcium sulfate, 65% β-tricalcium phosphate).
  Interventions: Procedure: Autogenous Bone Block + Xenograft + Collagen Membrane

INTERVENTIONS:
Procedure: Autogenous Bone Block + Xenograft + Collagen Membrane — Autogenous chin bone block graft combined with particulate bovine xenograft (Bio-Oss, Geistlich Pharma AG) and covered with an absorbable collagen membrane (Bio-Gide).

SUMMARY:
. Group A, received ABG cylinders obtained from the chin and organic bovine bone mineral particles (Bio-Oss xenograft) along with an absorbable collagen membrane. ABG cylinders from the chin and biphasic alloplastic (EthOss) grafting material made of CS (35%) and TCP (65%) were given to Group B. CBCT scans were conducted before bone augmentation surgery, one week and 6 months postoperatively

DETAILED DESCRIPTION:
Two groups of forty patients participated in this prospective, controlled, randomized clinical investigation. Group A, received ABG cylinders obtained from the chin and organic bovine bone mineral particles (Bio-Oss xenograft) along with an absorbable collagen membrane. ABG cylinders from the chin and biphasic alloplastic (EthOss) grafting material made of CS (35%) and TCP (65%) were given to Group B. CBCT scans were conducted before bone augmentation surgery, one week and 6 months postoperatively

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years requiring implant-supported restoration in the anterior maxilla

Horizontal alveolar bone deficiency <4 mm (Cawood & Howell Class III-IV)

Satisfactory oral hygiene

No previous bone augmentation at study site

Exclusion Criteria:

* Uncontrolled systemic diseases

History of head/neck irradiation or immunosuppression

Oral lesions (e.g., lichen planus)

Ongoing or recent IV bisphosphonate therapy

Untreated periodontitis or poor oral hygiene

Parafunctional habits, pregnancy, psychiatric disorders

Recent tobacco use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Change in horizontal alveolar ridge width | Baseline, 1 week, and 6 months post-surgery

SECONDARY OUTCOMES:
Postoperative complications | Up to 6 months post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine, Nahda University,Taibah University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No